CLINICAL TRIAL: NCT00569764
Title: The Effects of Metabolic Parameters of Aripiprazole in Patients With Schizophrenia
Brief Title: Effect on Metabolic Parameters of Abilify in SPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National Hospital (Other Government)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Jong-il Lee, Seoul National Hospital
Other Study IDs: snh002; MSABLI
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia; Metabolic Syndrome
Keywords: schizophrenia; metabolic syndrome; aripiprazole
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational: patients with schizophrenia who want to change an antipsychotics due to metabolic side effect

SUMMARY:
To measure the long-term changes in weight and plasma lipids after switching antipsychotic treatment to aripiprazole

DETAILED DESCRIPTION:
To measure the long-term changes in weight, plasma lipids and fasting blood glucose after switching antipsychotic treatment to aripiprazole, 1 year, open label studies in out and in-patients with schizophrenia.

The measurement of weight and lipid profile and fasting blood glucose will be measured at baseline and every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis with schizophrenia
* who signed an informed consent

Exclusion Criteria:

* comorbid with substance abuse or substance dependence
* pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with schizophrenia who want to change an antipsychotics due to metabolic side effects
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-12; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
weight lipid profile : HDL, LDL, total-cholesterol, triglyceride fasting blood glucose | 1 year

SECONDARY OUTCOMES:
prolactin ECG | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jong-il Lee, M.D., Study Director — Seoul National Hospital
Locations (1):
- Seoul National Hospital, Seoul, South Korea